CLINICAL TRIAL: NCT03794882
Title: Impact of Preoperative Quadratus Lumborum Block on Recovery Profile After Laparoscopic Ventral Hernia Repair
Brief Title: Impact of Quadratus Lumborum Block on Recovery Profile After Ventral Hernia Repair
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: administrative challenges and complications due to the COVID-19 pandemic
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018-0793; A530900 (Other: UW Madison); SMPH/ANESTHESIOLOGY/ANESTHESIO (Other: UW Madison); Protocol Version 8/26/2019 (Other: UW Madison)
Record Dates: First submitted 2018-12-20; First posted 2019-01-07 (Actual); Results first posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-08

CONDITIONS: Pain, Postoperative; Opioid Use
Keywords: Hernia, Ventral; Pain, Postoperative; Opioid Use; Pain
MeSH Terms: conditions — Pain, Postoperative; Hernia, Ventral; Pain

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: The participant is blinded to the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- QLB + Medical Management (Experimental): Subjects will undergo Intervention: Procedure/Surgery: Quadratus Lumborum Block and receive Intervention: Procedure: Standard Medical Management as needed.
  Interventions: Combination Product: Quadratus Lumborum Block; Procedure: Standard Medical Management
- Standard Medical Management (Active Comparator): Subjects will receive Intervention: Procedure: Standard Medical Management as needed.
  Interventions: Procedure: Standard Medical Management

INTERVENTIONS:
Combination Product: Quadratus Lumborum Block — 30 mL of .25% bupivacaine with 2.5mcg/mL epinephrine will be injected on both sides of the mid-abdomen posterior to the mid-axillary line.
  Other Names: QLB
  Arms: QLB + Medical Management
Procedure: Standard Medical Management — Standard medical management typically includes perioperative multimodal analgesia utilizing acetaminophen, opioids, non-steroidal anti-inflammatory drugs, and dexamethasone

SUMMARY:
Ventral hernia repair may be associated with significant postoperative pain. Pain is typically managed with intravenous (IV) and oral medications that come with their own risks, such as nausea, constipation, sedation, respiratory depression, increased bleeding, and/or kidney or liver dysfunction. The quadratus lumborum peripheral nerve block has been shown to produce anesthesia of the anterior abdominal wall in the T7 to L1 distribution. This study aims to evaluate if the addition of the quadratus lumborum peripheral nerve block (QLB) can improve pain scores, decrease the need for IV and oral pain medications, and/or speed the patients' return to normal activity.

DETAILED DESCRIPTION:
Current trends in perioperative pain management stress the importance of multimodal analgesia in an effort to reduce the dependence on opioid pain medications. Adverse effects of opioids include sedation, respiratory depression, nausea, vomiting, constipation, itching, and, most importantly, the potential for tolerance and abuse. Multimodal analgesia attempts to utilize multiple techniques, including medications and nerve block procedures, to improve postoperative analgesia. Improved postoperative pain control can enable an earlier return to normal activities for patients, not only improving patient satisfaction, but also reducing postoperative morbidity and adverse effects of opioids.

Approximately 350,000 to 500,000 ventral hernia repairs are performed each year in the United States. Surgeries completed laparoscopically are typically performed on an outpatient basis, allowing patients to return home the same day of surgery and treat their pain independently with prescribed pain medications. Utilization of a regional anesthesia technique may allow prolonged numbing of the nerves postoperatively and decrease the reliance on oral pain medications. Transversus abdominis plane (TAP) blocks have been shown to decrease pain scores and opioid consumption following ventral hernia repair. Quadratus lumborum (QL) blocks are newer iterations of the TAP block.

There are currently three types of the QL block, all targeting the thoracolumbar fascia surrounding the quadratus lumborum muscle. Injection within this fascial plane may allow local anesthetic spread into the paravertebral space, possibly explaining why QL blocks have been mapped from the T7 to T12/L1 dermatomes, covering the entire abdomen. Conversely, TAP blocks have been mapped from the T10 to T12/L1 dermatomes, only covering the abdomen below the umbilicus. In the first, the Quadratus lumborum 1 block (QL1), the local anesthetic is injected within the fascial plane lateral to the QL muscle. In the second, the Quadratus lumborum 2 block (QL2), the needle trajectory is more superficial, and the local anesthetic is injected along the posterior border of the QL muscle. The third iteration, the Quadratus lumborum 3 block (QL3), involves a deeper, transmuscular approach with injection along the anterior border of the QL muscle. Our study would utilize the QL2 approach as the dermatomal distribution of the QL1 and QL2 blocks appear to be more widespread than the QL3 block, and the QL2 block may be a safer approach due to the more superficial angle of the needle 3.

Additionally, the QL block has been shown to have a longer duration of analgesia when directly compared to the TAP block. A study of pediatric lower abdominal surgery revealed improved pain scores and parent satisfaction with care in the QL group compared to TAP block. This improvement persisted to the 24 hour mark. In a study of postoperative pain following cesarean delivery, pain scores were improved and opioid consumption decreased with the QL block compared to the TAP block. The differences were not significant at the 1 and 6 hour marks, but were significant at the 12, 24 and 48 hour marks, highlighting the analgesic duration of the QL block 8.

This study aims to evaluate the efficacy of the QL block using the QL2 approach on recovery profile after laparoscopic ventral hernia repair, a commonly performed surgery, as well as contribute to the understanding of the block and its distribution of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is scheduled for elective laparoscopic ventral hernia repair;
2. The subject is ≥ 18 years and ≤ 80 years;
3. The patient agrees to receive a quadratus lumborum block
4. American Society of Anesthesiologists class 1-3.

Exclusion Criteria:

1. Subject is < 18 years of age or >80 years of age;
2. Subject is non-English speaking;
3. Subject is known or believed to be pregnant;
4. Subject is a prisoner;
5. Subject has impaired decision-making capacity per discretion of the Investigator;
6. Significant renal, cardiac or hepatic disease per discretion of the investigator;
7. American Society of Anesthesiologists class 4-5;
8. Known hypersensitivity and/or allergies to local anesthetics;
9. Chronic opioid use (daily or almost daily use of opioids for > 3 months at any point in their lives).
10. Repair of a recurrent ventral hernia
11. Repair of multiple ventral hernias
12. Unobtainable sonographic views
13. Lacking health insurance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Bevil, MD, Principal Investigator — Anesthesiology Department, University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States,53792.
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- QLB + Medical Management: Subjects will undergo Intervention: Procedure/Surgery: Quadratus Lumborum Block and receive Intervention: Procedure: Standard Medical Management as needed.
  Quadratus Lumborum Block: 30 mL of .25% bupivacaine with 2.5mcg/mL epinephrine will ne injected on both sides of the mid-abdomen posterior to the mid-axillary line.
  Standard Medical Management: Standard medical management typically includes perioperative multimodal analgesia utilizing acetaminophen, opioids, non-steroidal anti-inflammatory drugs, and dexamethasone
Period: Overall Study
Arm/Group | QLB + Medical Management | Standard Medical Management
Started | 8 | 6
Completed | 8 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QLB + Medical Management | Standard Medical Management | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Continuous [Mean (Full Range); unit: years] | 49.38 [25 to 68] | 56.17 [40 to 67] | 54.69 [25 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 8 | 6 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Day (POD) 1 Pain Score
Description: Pain Score assessed on POD 1 using a Numerical Rating Scale (NRS) (0-10) where 0 represents no pain and 10 represents the worst pain imaginable.
Time Frame: 24 hours
Population: Not all participants answered the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QLB + Medical Management | Standard Medical Management
Number analyzed (Participants) | 8 | 5
score on a scale | 3.7857 (1.643) | 4.015 (2.291)

2. Secondary Outcome: Pain Score at Rest
Description: Pain at rest in PACU, and on POD 1, 2, 7 using a Numerical Rating Scale (NRS) (0-10) where 0 represents no pain and 10 represents the worst pain imaginable.
Time Frame: PACU, POD1, POD2, POD7
Population: Not all participants answered the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QLB + Medical Management | Standard Medical Management
Number analyzed (Participants) | 8 | 6
score on a scale
  Pain Score at Rest PACU | 7.5833 (2.224) | 7.12 (1.443)
  Pain at Rest POD 1: number analyzed (Participants) | 7 | 6
  Pain at Rest POD 1 | 3.88 (1.64) | 3.50 (2.25)
  Pain at Rest POD 2: number analyzed (Participants) | 6 | 6
  Pain at Rest POD 2 | 3.33 (0.96) | 3.00 (1.73)
  Pain at Rest POD 7: number analyzed (Participants) | 7 | 6
  Pain at Rest POD 7 | 1.43 (1.03) | 1.57 (1.34)

3. Secondary Outcome: Pain Score With Activity
Description: Pain with activity in PACU and on POD 1, 2, 7 assessed using a Numerical Rating Scale (NRS) (0-10) where 0 represents no pain and 10 represents the worst pain imaginable.
Time Frame: PACU, POD1, POD2, POD7
Population: Not all participants answered survey questions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QLB + Medical Management | Standard Medical Management
Number analyzed (Participants) | 8 | 6
score on a scale
  Pain Score with Activity PACU: number analyzed (Participants) | 0 | 0
  Pain Score with Activity POD 1: number analyzed (Participants) | 7 | 6
  Pain Score with Activity POD 1 | 7.07 (2.20) | 6.75 (1.97)
  Pain Score with Activity POD 2: number analyzed (Participants) | 6 | 6
  Pain Score with Activity POD 2 | 7.00 (2.57) | 5.58 (1.41)
  Pain Score with Activity POD 7: number analyzed (Participants) | 7 | 6
  Pain Score with Activity POD 7 | 3.5712 (2.012) | 3.670 (1.155)

4. Secondary Outcome: Opioid Consumption in Oral Morphine Milligram Equivalent (OMME)
Description: Opioid Consumption in morphine equivalents in PACU and on POD, 1, 2, 7.
Time Frame: PACU, POD1, POD2, POD7
Population: 3 participants from the QLB + Management Group did not respond to the 7 day OMME question.
Measure: Mean (Standard Deviation); unit: OMME
Arm/Group | QLB + Medical Management | Standard Medical Management
Number analyzed (Participants) | 5 | 6
OMME
  Opioid Consumption in PACU | 28.93 (25.65) | 36.64 (16.70)
  Opioid Consumption POD 1 | 24.58 (15.31) | 19.50 (2.89)
  Opioid Consumption POD 2 | 27.50 (17.00) | 20.50 (5.77)
  Opioid Consumption POD 7 | 58 (79.88) | 66.5 (37.27)

5. Secondary Outcome: Location of Most Severe Pain
Description: Location of most severe pain on assessed by questioning the patient in PACU and on POD 1, 2, 7.
Time Frame: PACU, POD1, POD2, POD7
Population: Two subjects on the expermental protocol and one in the control group were unable to provide the answers to this secondary aim question when asked by the study team.
Measure: Count of Participants; unit: Participants
Arm/Group | QLB + Medical Management | Standard Medical Management
Number analyzed (Participants) | 8 | 6
Participants
  PACU: number analyzed (Participants) | 6 | 5
  PACU: around navel | 4 | 2
  PACU: incision area | 2 | 2
  PACU: abdomen | 0 | 0
  PACU: navel | 0 | 1
  PACU: stomach area | 0 | 0
  PACU: middle of abomen | 0 | 0
  PACU: middle | 0 | 0
  POD 1: number analyzed (Participants) | 7 | 4
  POD 1: around navel | 0 | 0
  POD 1: incision area | 2 | 2
  POD 1: abdomen | 2 | 2
  POD 1: navel | 0 | 0
  POD 1: stomach area | 1 | 0
  POD 1: middle of abomen | 1 | 0
  POD 1: middle | 1 | 0
  POD 2: number analyzed (Participants) | 7 | 6
  POD 2: around navel | 1 | 1
  POD 2: incision area | 3 | 2
  POD 2: abdomen | 1 | 2
  POD 2: navel | 0 | 0
  POD 2: stomach area | 0 | 1
  POD 2: middle of abomen | 2 | 0
  POD 2: middle | 0 | 0
  POD 7: number analyzed (Participants) | 5 | 5
  POD 7: around navel | 0 | 0
  POD 7: incision area | 3 | 2
  POD 7: abdomen | 0 | 2
  POD 7: navel | 0 | 1
  POD 7: stomach area | 2 | 0
  POD 7: middle of abomen | 0 | 0
  POD 7: middle | 0 | 0

6. Secondary Outcome: Time in PACU
Description: Duration of patients' time in PACU.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | QLB + Medical Management | Standard Medical Management
Number analyzed (Participants) | 8 | 6
minutes | 66.63 (28.58) | 64.33 (26.82)

7. Secondary Outcome: Postoperative Time to Discharge
Description: Total postoperative time until discharge.
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | QLB + Medical Management | Standard Medical Management
Number analyzed (Participants) | 8 | 5
hours | 66.625 (28.58) | 66.60 (26.82)

8. Secondary Outcome: Numbness Distribution in PACU
Description: For patients that underwent QLB, numbness to ice will be assessed by filling a plastic glove with ice water and systematically assessing numbness to cold in the thoracic and lumbar dermatomes by comparing these sites with a reference point.
Time Frame: 12 hours
Population: This question was not asked by the clinical team at 12 hours and therefore, no data can be entered for this aim.
Arm/Group | QLB + Medical Management | Standard Medical Management
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants Who Report Nausea in PACU
Description: Patient will be questioned to assess if they have nausea in PACU.
Time Frame: 12 hours
Measure: Count of Participants; unit: Participants
Arm/Group | QLB + Medical Management | Standard Medical Management
Number analyzed (Participants) | 8 | 5
Participants | 2 | 0

10. Secondary Outcome: Total Antiemetic Consumption on POD 0 and in PACU
Description: Total consumption of antiemetics on POD 0 and in PACU.
Time Frame: 12 hours
Population: This secondary aim was not asked/followed up by the PI and therefore, the subjects were not asked this question and no data was collected for either time point.
Arm/Group | QLB + Medical Management | Standard Medical Management
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Participants With Presence of Nausea Necessitating Treatment
Description: Patient will be questioned to assess if they had nausea necessitating treatment on POD 1, 2, and 7
Time Frame: POD1, POD2, POD7
Population: Data was not collected from all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | QLB + Medical Management | Standard Medical Management
Number analyzed (Participants) | 5 | 4
Participants
  POD 1 | 5 | 4
  POD 2 | 0 | 0
  POD 7 | 0 | 0

12. Secondary Outcome: Rating of Satisfaction With Perioperative Care
Description: Satisfaction with perioperative care on POD 1, 2, and 7 measured by a Numerical Rating Scale (0-10) with 0 representing no satisfaction and 10 representing high satisfaction.
Time Frame: POD1, POD2, POD7
Population: Not all participants responded to the survey question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QLB + Medical Management | Standard Medical Management
Number analyzed (Participants) | 7 | 5
score on a scale
  Rating of Satisfaction with perioperative care POD 1 | 8.60 (0.97) | 9.20 (1.14)
  Rating of Satisfaction with perioperative care POD 2 | 8.83 (0.96) | 9.17 (1.91)
  Rating of Satisfaction with perioperative care POD 7 | 9.21 (1.096) | 8.61 (1.768)

13. Secondary Outcome: Total Non-Opioid Analgesic Consumption in PACU: Measured in Milligrams
Description: Total consumption of Non-Opioid Analgesics in the PACU.
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | QLB + Medical Management | Standard Medical Management
Number analyzed (Participants) | 8 | 6
milligrams
  Ketorolac | 0 (0) | 5 (12.25)
  lidocaine in mg | 0 (0) | 0 (0)
  acetaminophen in mg | 235.71 (415.04) | 333.33 (440.17)

14. Secondary Outcome: Additional Analgesics in Milliliters Administered in the Operating Room
Description: This measure describes the amount, in milliliters, of non-opioid analgesics administered in the Operating Room.
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | QLB + Medical Management | Standard Medical Management
Number analyzed (Participants) | 8 | 6
milliliters | 0 (0) | 15.00 (16.43)

15. Secondary Outcome: Additional Analgesics in Milligrams Administered in the Operating Room
Description: This measure describes the amount, in milligrams, of non-opioid analgesics administered in the Operating Room.
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | QLB + Medical Management | Standard Medical Management
Number analyzed (Participants) | 8 | 6
milligrams
  Ketorolac | 8.57 (8.02) | 2.50 (6.12)
  Acetaminophen | 166.67 (408.25) | 0 (0)
  Propofol | 0.00 (0.00) | 28.33 (69.40)
  lidocaine | 17.50 (36.15) | 20.00 (40.00)

ADVERSE EVENTS:
Time Frame: up to Post-operative day 7 (POD7)
Arm/Group | QLB + Medical Management | Standard Medical Management
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/8 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QLB + Medical Management (N=8) | Standard Medical Management (N=6)
incision site bleeding (General disorders) | 0 (0) | 1 (1) — The subject reported incision site bleeding and tiredness at the 7 day time period.
tiredness (General disorders) | 0 (0) | 1 (1) — Overall tiredness

LIMITATIONS AND CAVEATS:
This study was terminated early due to the combined effects of the COVID-19 pandemic and the switching of the primary location for the procedure from UW Hospital to East Madison Hospital.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/82/NCT03794882/Prot_SAP_000.pdf